CLINICAL TRIAL: NCT00149695
Title: Soft Drink, Milk and Obesity in Chilean Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Charles H. Hood Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TW006818-Fogarty (completed); R03TW006818 (NIH)
Record Dates: First submitted 2005-08-31; First posted 2005-09-08 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Obesity
Keywords: Obesity, beverages, weight loss, body mass index, diet
MeSH Terms: conditions — Obesity; Weight Loss

INTERVENTIONS:
Behavioral: Weekly home delivery of milk products

SUMMARY:
The primary aim of this randomized controlled trial is to evaluate the effects of replacing habitual consumption of sugar-sweetened soft drinks with milk over 16 weeks.

DETAILED DESCRIPTION:
The prevalence of obesity has risen dramatically among children in the U.S. and throughout the world since the 1960s. Many factors are thought to have contributed to the epidemic of pediatric obesity. One factor that has received increasing attention is consumption of sugar-sweetened beverages. Feeding studies suggest physiological mechanisms by which sugar in liquid form may be less satiating than other foods. An observational study found total energy consumption to be greater among children who consume sugar-sweetened beverages compared to non-consumes. Short-term interventional studies report increasing energy intake and body weight in subjects given sugar-sweetened beverages compared to non-caloric beverages. Our preliminary data found that the risk for becoming obese increased by about 60% in middle school children for every additional serving per day of sugar-sweetened beverage consumed. The purpose of the present study is to conduct a 16-week clinical trial involving 96 children ages 8 to 10 years in Chile, a developing nation characterized as undergoing a "nutrition transition." The subjects, selected for current sugar-sweetened soft drink consumption, will be randomly assigned to intervention or control groups. The intervention group will be encouraged to substitute milk products for soft-drinks; to facilitate this dietary change, a variety of milk products will be delivered to subjects' homes on a weekly basis. Clinical endpoints include changes in dietary quality, body weight, adiposity by DEXA-scan and measures of calcium homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 8 to 10 years
* Tanner Stage I
* BMI between 85th and 95th percentiles for age and gender
* Consuming at least 2 servings/day of sugar-sweetened beverages
* Willingness to consume milk instead of sugar-sweetened beverages for 16 weeks
* Able to read Spanish and accurately complete dietary assessments

Exclusion Criteria:

* Presence of a serious underlying medical condition
* Taking any medication that affects body weight
* History of lactose intolerance or milk protein allergies
* History of an eating disorder

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96
Dates: Start 2004-07; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change in percent body fat by DXA scan

SECONDARY OUTCOMES:
Body mass index
Blood glucose
Blood insulin
Serum lipids

CONTACTS AND LOCATIONS:
Overall Officials: David S Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital; Cecilia Albala, MD, Principal Investigator — INTA - University of Chile; Cara B Ebbeling, PhD, Study Director — Boston Children's Hospital; Mariana Cifuentes, PhD, Study Director — INTA - University of Chile
Locations (1):
- INTA - University of Chile, Santiago, Chile

REFERENCES:
- [Background] Ludwig DS, Peterson KE, Gortmaker SL. Relation between consumption of sugar-sweetened drinks and childhood obesity: a prospective, observational analysis. Lancet. 2001 Feb 17;357(9255):505-8. doi: 10.1016/S0140-6736(00)04041-1. PMID 11229668
- [Background] Pereira MA, Jacobs DR Jr, Van Horn L, Slattery ML, Kartashov AI, Ludwig DS. Dairy consumption, obesity, and the insulin resistance syndrome in young adults: the CARDIA Study. JAMA. 2002 Apr 24;287(16):2081-9. doi: 10.1001/jama.287.16.2081. PMID 11966382
- [Derived] Albala C, Ebbeling CB, Cifuentes M, Lera L, Bustos N, Ludwig DS. Effects of replacing the habitual consumption of sugar-sweetened beverages with milk in Chilean children. Am J Clin Nutr. 2008 Sep;88(3):605-11. doi: 10.1093/ajcn/88.3.605. PMID 18779274